CLINICAL TRIAL: NCT02702336
Title: EYTO-kids: European Youth Tackling Obesity in Adolescents and Children, Una intervención Para Mejorar Los Estilos de Vida (Estudio Piloto)
Brief Title: EYTO-kids-Pilot: European Youth Tackling Obesity in Adolescents and Children.
Acronym: EYTO-kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Rosa Sola, Full Professor, MD, PhD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EYTO-Kids-Pilot
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Dietary Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EYTO-Kids Intervention Group (Experimental): Adolescents will receive 16h of training (2h healthy lifestyle training, social marketing and communication, 6h to design activities, 2h session together with all intervention high-schools, 6h to practice and standardize activities) and 4h (1h/activity) to implement 4 activities in schools. The scholars will receive 4 activities designed by adolescents, focusing on: 1) increasing fruit consumption, 2) increasing vegetable consumption, 3) increasing physical activity practice and to reduce sedentary lifestyles and, 4) decreasing sugary drinks and fast-food consumption.
  Interventions: Behavioral: EYTO-kids
- Control Group (No Intervention): The control group will not receive any kind of intervention (only the assessment).

INTERVENTIONS:
Behavioral: EYTO-kids — To promote healthy lifestyles among young people, through the design and implementation of health promotion activities carried out by adolescents (12-14 years old) to scholars of primary education (8-10 years old), using social marketing and peer-led strategy.
  Arms: EYTO-Kids Intervention Group

SUMMARY:
The primary aim is to promote healthy lifestyles among young people, through the design and implementation of health promotion activities carried out by adolescents (12-14 years old) to scholars of primary education (8-10 years old), using social marketing and peer-led strategy.

The secondary aims are: 1) to increase fruit and vegetable consumption and physical activity practice in scholars and adolescents; 2) to reduce sedentary lifestyles, sugary drinks and fast-food in scholars and adolescents.

The EYTO-kids program is a randomized, parallel, intervention program with control group, with a 2 academic courses, 2015-2016 to 2016-2017 (10 months in total), in Reus (Spain).

To achieve the aims, social marketing and peer-led methodologies will be used at the intervention design and implementation. Adolescents from secondary education (1st /2nd ESO: Educación Secundaria Obligatoria-Obligatory Secondary Education) will design and implement activities to scholars from primary education (3rd/4th primary education).

The adolescents from the intervention group will design and implement activities to implement them in to children, and the control group will not receive any kind of intervention (only the assessment).

Participation will occur according to the randomized sample size, where a minimum of 208 adolescents (104 as intervention and 104 as control group), and 602 scholars (301 as intervention and 301 as control group) will be involved.

The inclusion criteria are: to have signed informed consent (from mother/father/guardian of the participant), to provide basic demographic data, to assist participating schools and to answer a lifestyle questionnaire.

DETAILED DESCRIPTION:
Nowadays, unhealthy lifestyles are associated with some chronic diseases, especially obesity. If the improvement of healthy lifestyles occurs during childhood or adolescence, long-term effectiveness can be achieved. To improve healthy lifestyles, interventions that use strategies such as social marketing (based on commercial marketing, including 8 criteria to choice healthy options) and peer-led methodology (also known as peer education, is based in the transmission of healthy messages from peers to peers), have demonstrated effectiveness in youth health promotion.

The primary aim is to promote healthy lifestyles among young people, through the design and implementation of health promotion activities carried out by adolescents (12-14 years old) to scholars of primary education (8-10 years old), using social marketing and peer-led strategy.

The secondary aims are: 1) to increase fruit and vegetable consumption and physical activity practice in scholars and adolescents; 2) to reduce sedentary lifestyles, sugary drinks and fast-food in scholars and adolescents.

The EYTO-kids program is a pilot cluster, randomized, parallel, intervention program with control group, with a 2 academic courses, 2015-2016 to 2016-2017 (10 months in total), in Reus (Spain).

To achieve the aims, social marketing and peer-led methodologies will be used at the intervention design and implementation. Adolescents from secondary education (1st /2nd ESO: Educación Secundaria Obligatoria-Obligatory Secondary Education) will design and implement activities to scholars from primary education (3rd/4th primary education).

The adolescents from the intervention group will design and implement activities to implement them in to children, and the control group will not receive any kind of intervention (only the assessment).

Participation will occur according to the randomized sample size, where a minimum of 208 adolescents (104 as intervention and 104 as control group), and 602 scholars (301 as intervention and 301 as control group) will be involved.

The inclusion criteria are: to have signed informed consent (from mother/father/guardian of the participant), to provide basic demographic data, to assist participating schools and to answer a lifestyle questionnaire.

The intervention:

Adolescents will receive 16h of training (2h healthy lifestyle training, social marketing and communication, 6h to design activities, 2h session together with all intervention high-schools, 6h to practice and standardize activities) and 4h (1h/activity) to implement 4 activities in schools.

The scholars will receive 4 activities designed by adolescents, focusing on: 1) increasing fruit consumption, 2) increasing vegetable consumption, 3) increasing physical activity practice and to reduce sedentary lifestyles and, 4) decreasing sugary drinks and fast-food consumption.

All participants (intervention and control group) will respond a questionnaire composed by 4 validated questionnaires (ENkid questionnaire, AVall questionnaire, HBSC questionnaire and HABITS questionnaire).

It is expected to increase the percentage of scholars and adolescents that:

Consume 1 fruit/day (primary outcome) Consume 1 vegetable/day

Practice ≥4h/week physical activity practice (primary outcome)

And decrease the percentage of scholars and adolescents that:

Practice sedentary lifestyles Consume sugary drinks every day Attend ≥ once/week to fast-food restaurants.

ELIGIBILITY:
Inclusion Criteria:

* to have signed informed consent (from mother/father/guardian of the participant)
* to provide basic demographic data
* to assist participating schools and,
* to answer a lifestyle questionnaire.

Exclusion Criteria:

* Lack of one of the inclusion criteria.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 810 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Fruit consumption and Physical Activity practice | 10 months
  Increase ≥1/day fruit consumption; Increase ≥4h/week physical activity practice

SECONDARY OUTCOMES:
Vegetable consumption | 10 months
  Consume ≥1 vegetable/day
Sugary Drinks | 10 months
  Reduce sugary drinks every day
Fast-food | 10 months
  Decrease to attend ≥ once/week to fast-food restaurants.
Sedentary behaviours practice | 10 months
  Decrease sedentary behaviours practice

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, MD, PhD, Principal Investigator — University Rovira i Virgili

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Bell SL, Audrey S, Cooper AR, Noble S, Campbell R. Lessons from a peer-led obesity prevention programme in English schools. Health Promot Int. 2017 Apr 1;32(2):250-259. doi: 10.1093/heapro/dau008. PMID 24711350
- [Derived] Tarro L, Llaurado E, Aceves-Martins M, Morina D, Papell-Garcia I, Arola L, Giralt M, Sola R. Impact of a youth-led social marketing intervention run by adolescents to encourage healthy lifestyles among younger school peers (EYTO-Kids project): a parallel-cluster randomised controlled pilot study. J Epidemiol Community Health. 2019 Apr;73(4):324-333. doi: 10.1136/jech-2017-210163. Epub 2019 Jan 25. PMID 30683803